CLINICAL TRIAL: NCT07180654
Title: Pilot Study on Menstrual Cycle-Related Hormonal Effects on Motor Cortex Plasticity Assessed by TMS in Healthy Young Adults
Brief Title: Menstrual Cycle TMS Plasticity Pilot
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 858764
Record Dates: First submitted 2025-09-02; First posted 2025-09-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cortical Activation
Keywords: transcranial magnetic stimulation; cortical excitability; hormones
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Participants may be asked to provide blood samples. This analysis may measure serum estradiol, progesterone, testosterone, luteinizing hormone, and/or follicle-stimulating hormone. No more than 10 mL of blood may be collected at each visit. Blood will be collected at Penn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Volunteers: Single group design
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Subjects will receive a series of 60 10s trains that will be presented over the course of the ~3.5 min session. Each train will consist of 2 s of stimulation with an 8 s ITI. During the 2 s of stimulation, 10, 50 Hz bursts will be repeated at intervals of 200 ms (5 Hz). iTBS will be administered at 100% of the motor threshold (MT).

SUMMARY:
Aim 1: Assess how menstrual cycle phase affects motor cortex plasticity in females.

Aim 2: Compare motor cortex plasticity between males and females across the same time points, identifying potential sex differences in TMS response.

Aim 3: Examine associations between serum hormone levels and TMS-induced plasticity within and between sexes.

DETAILED DESCRIPTION:
This project will recruit healthy male and female volunteers between the ages of 20-40. Females must who are not on hormonal medications and, if female, have regular menstrual cycles as defined in Table 1. At time of consent, female participants will be send home with given tests that may assess urine estradiol, LH and/or their metabolites. Participants will be asked to complete these tests at home, will be instructed to use these tests in the morning at the first void of the day; the number of days during each cycle that participants will be asked to complete these tests will be based on their report of their regular cycle pattern but will not be longer than half the number of days in each cycle. In addition, female subjects will be given a RedCap survey link at which they will track their menstrual cycle and results from the urine estradiol/LH tests.

Subjects will undergo 4 study visits over approximately 1-2 months depending on availability and, if female, menstrual cycle point. At visit 1, subjects will consent to the protocol, fill out surveys including the TMS Adult Safety Screening (TASS) and a questionnaire about past hormonal medication use and if relevant, menstrual cycle history. If female, subjects will be given take-home ovulation tests to use across the study duration.

On the following visits, they may undergo the following procedures: 1) venipuncture to collect approximately 45mL 10 mL of blood 2) motor threshold testing, 2) Paired-Pulse Stimulation 3) Single-Pulse TMS to the motor cortex 4) intermittent Theta Burst Stimulation (iTBS) to the motor cortex.

ELIGIBILITY:
Inclusion Criteria:

* Able to give their consent
* If female, must have menstrual cycles of normal frequency, regularity, and duration.

Exclusion Criteria:

* Non-English speaking
* Any medical condition that increases risk for TMS
* History of seizure
* History of epilepsy
* Increased risk of seizure for any reason

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the community in the Philadelphia Metro Area.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Single-pulse TMS | Will be collected during 3 visits over the course of a 2 month timeframe during different phases of the menstrual cycle (in females).
  Single-pulse TMS: Cortical excitability curves will be measured before and after a single 1800-pulse train of iTBS. Motor Evoked Potentials (MEPs) will be recorded from the right FDI muscle at 7 distinct intensities ranging from -20% to + 40% of MT. Single pulses will be delivered once every 10±3 seconds to the left motor cortex at random intensities in the above range to avoid habituation across pulses. Across the session, a total of 70 pulses will be delivered before and after iTBS, 10 at each intensity.
Paired pulse stimulation | Will be collected during 3 visits over the course of a 2 month timeframe during different phases of the menstrual cycle (in females).
  Paired-pulse stimulation: Subjects will undergo paired-pulse stimulation to measure both intracortical inhibition and intracortical facilitation. For intracortical inhibition, subjects will receive a conditioning pulse at 80% MT 4 seconds before the test pulse at 120% MT. For intracortical facilitation, subjects will receive a conditioning pulse at 120% MT 15s before the test pulse at 120% MT. Across the session, a total of 60 paired pulses will be delivered before and after iTBS, 30 at each ISI.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Balderston, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided